CLINICAL TRIAL: NCT03980288
Title: A Phase I Clinical Study of 4th Generation Chimeric Antigen Receptor T Cells Targeting Glypican-3 ( CAR-GPC3 T Cells) in Patients With Advanced Hepatocellular Carcinoma
Brief Title: 4th Generation Chimeric Antigen Receptor T Cells Targeting Glypican-3
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: CARsgen Therapeutics Co., Ltd. (Industry)
Responsible Party: Principal Investigator, TingBo Liang, Professor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CISLD-4
Record Dates: First submitted 2019-06-02; First posted 2019-06-10 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Advanced Hepatocellular Carcinoma
Keywords: Advanced hepatocellular Carcinoma; CAR-T; GPC3

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-GPC3 T Cells (Experimental): The subjects enrolled will be sequentially assigned to Part 1 at 3 dose levels via typical 3+3 dose escalation method and then Part 2, cohort expansion stage, 3 cohorts of CAR T therapy combination with currently available treatment for HCC. stage Part 1: Dose escalating: 3 dose level Part 2: 3 cohorts Cohort 1. Combination with tyrosine kinase inhibitors Cohort 2. Combination with PD-1 / PD-L1 monoclonal antibody Cohort 3. Combination with the drugs may benefit for patient at investigator's discretion
  Interventions: Drug: CAR-GPC3 T Cells

INTERVENTIONS:
Drug: CAR-GPC3 T Cells — Pretreatment with fludarabine and cyclophosphamide CAR-GPC3 T Cells infusion

SUMMARY:
A Phase I Clinical Study of 4th generation Chimeric Antigen Receptor T Cells Targeting Glypican-3 ( CAR-GPC3 T Cells) in Patients with Advanced Hepatocellular Carcinoma

DETAILED DESCRIPTION:
This is a phase I open-label, single and multiple infusion, dose escalation/cohort expansion study to evaluate the safety, cell pharmacokinetics, and preliminary efficacy of CAR-GPC3 T cells, infused intravenously in subjects who have been diagnosed with GPC3 positive advanced hepatocellular carcinoma and refractory or intolerant to current standard systemic treatment.

Primary objectives:

•To evaluate the safety and tolerability of CAR-GPC3 T cells infused intravenously at escalating doses in patients with advanced hepatocellular carcinoma.

Secondary objectives:

* To evaluate the cellular pharmacokinetics of CAR-GPC3 T cells
* To evaluate the overall safety and tolerability of infusion of CAR-GPC3 T cells
* To investigate the preliminary efficacy of CAR-GPC3 T cells in the treatment of advanced hepatocellular carcinoma

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 75 years, male or female;
2. Patients with advanced hepatocellular carcinoma (HCC) diagnosed by histopathology or cytology who are not suitable for surgery or local treatment, have developed progressive disease or intolerability after standard systemic therapies (including but not limited to systemic chemotherapy, molecular targeted therapy);
3. According to BCLC, the patients are classified into Grade C or Grade B unsuitable for local treatment/progressive disease after local treatment;
4. In tumor tissue samples GPC3 is detected positive by immunohistochemistry (IHC);
5. According to RECIST 1.1, patients have at least one evaluable target lesion, defined as: the longest diameter of non-lymph node lesion ≥ 10 mm, or the shortest diameter of lymph node lesion ≥ 15 mm); hepatic lesions require arterial phase contrast enhancement;
6. Expected survival is > 12 weeks;
7. Cirrhosis status Child-Pugh score:≤7;
8. ECOG Performance Status score: 0 to 1 point;
9. If the patient is HBsAg positive or HBcAb positive, HBV-DNA should be <200 IU/ml. HBsAg positive patients must receive antiviral treatment according to the 2015 China Edition of Guideline for Chronic Hepatitis B Prevention and Treatment;
10. Subjects should have adequate organ functions before screening and pre-treatment (at baseline);
11. Have venous accesses for pheresis;
12. Subjects of childbearing age must undergo a serum pregnancy test within 14 days before the initiation of the study and the result must be negative. In addition, they should be willing to use a reliable method of contraception during the trial (within 52 weeks after cell infusion); male subjects whose spouses are women of childbearing age should undergo sterilization surgery or agree to use a reliable method of contraception during the trial;
13. Understand and sign informed consent.

Exclusion Criteria:

1. Pregnant or breast-feeding women;
2. HCV-RNA, HIV antibodies or Syphilis Serological tests are positive;
3. Any uncontrollable active infection, including but not limited to active tuberculosis;
4. Subjects have clinically significant thyroid dysfunction determined by investigator (serum thyroid hormone assays TT4, TT3, FT3, FT4, and serum thyroid stimulating hormone TSH) which is not suitable for entering into the study;
5. Previous or present hepatic encephalopathy;
6. Current clinically significant ascites, which is defined as ascites that are physically positive or require intervention (e.g., puncture or medication) for control (those whose imaging result shows ascites requiring no intervention may be included);
7. Imaging results:≥50% of the liver is replaced by tumor or portal vein main tumor thrombus, or tumor thrombus invasion of mesenteric vein / inferior vena cava;
8. Patients with known active autoimmune diseases which require to be treated with immunosuppressive agents including biological agents;
9. The side effects caused by the previous treatment of the subjects did not return to CTCAE ≤1; except hair loss and other tolerable events determined by investigator;
10. Patients who had received systemic steroids or other immunosuppressive agents within 2 weeks before collection of mononuclear cells, except those who had recently used or are currently using inhaled steroids;
11. Allergic to immunotherapy and related drugs;
12. Subjects have untreated or symptomatic brain metastases;
13. Subjects have central or extensively metastases in lung;
14. Subjects with unstable or active ulcers and gastrointestinal bleeding currently;
15. Patients with a history of organ transplantation or waiting for organ transplantation (including liver transplantation);
16. Subjects who have undergone antitumor therapy within 2 weeks prior to apheresis;
17. Previously received any chimeric antigen receptor-modified T-cells (CAR-T) , TCR T immunotherapy;
18. Subjects who have undergone PD-1/PD-L1 therapy within 3 months prior to screening;
19. Subjects who have undergone major surgery or significant trauma within 4 weeks prior to apheresis, or who are expected to undergo major surgery during the study;
20. There are no other serious diseases that may limit subjects' participation in this trial;
21. Prior to pretreatment and infusion,the subject has a central nervous system disease sign or an abnormal neurological test result with clinical significance;
22. Prior to pretreatment, subjects developed, including but not limited to, new arrhythmias that could not be controlled with drugs, hypotension requiring pressor agent, bacterial, fungal or viral infections that required intravenous antibiotics. Creatinine clearance rate <50mL/min; The investigator judges that the subject is not suitable for continuing the trial. Subjects who use antibiotics to prevent infection can continue the trials if judged by the investigator;
23. According to the investigators' evaluation, patients are unable or unwilling to comply with the requirements of the study protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-07-23 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Dose limited toxicity and Maximum Tolerated Dose | After 28 days of single infusion
  Safety and tolerability

SECONDARY OUTCOMES:
Number of cells | Through week 52 or the second timepoint of cells undetectable
  1.the number of cell copies and cell persistence duration in peripheral blood) Pharmacokinetics is the "Implantation endpoint" which is defined as the number of copies of the CAR-GPC3 DNA in peripheral blood detected at each visit after infusion until any two consecutive test results are negative or below the detection limit. Duration of CAR-GPC3 T Cell persistence is the period from the day of infusion to the first negative test result or result lower than the detection limit
Number of participants with treatment-related adverse events | Through study completion, an average of 3 years
  Adverse events occurring through18 weeks and 52weeks post infusion, such as abnormalities or changes in laboratory examinations, physical examinations, vital signs, etc.
  Adverse events occurring through18 weeks and 52weeks post infusion, such as abnormalities or changes in laboratory examinations, physical examinations, vital signs, etc.
Antitumor efficacy-Progression-free survival (PFS) | Through study completion, an average of 3 years
  The period from the day when the subject receives the first study treatment to the first recorded tumor progression (whether treated or not) or death of any cause, which occurs first
Antitumor efficacy-Duration of response (DOR) | Through study completion, an average of 3 years
  The period from the first evaluation of CR or PR to the first evaluation of PD or death of any cause.
Antitumor efficacy-Duration of disease control (DDC) | Through study completion, an average of 3 years
  The period from the first evaluation of CR, PR, or SD to the first evaluation of PD or any cause of death
Antitumor efficacy-Overall survival (OS) | Through study completion, an average of 3 years
  The period from the first study treatment to any cause of death
Antitumor efficacy-Objective response rate (ORR) | Through study completion, an average of 3 years
  The number of cases in which tumor size is reduced to PR or CR / the total number of evaluable cases (%). In the event of PR or CR, the subjects should confirm it no less than 4 weeks after the first evaluation
Antitumor efficacy-Disease control rate (DCR) | Through study completion, an average of 3 years
  The number of cases in which response (PR + CR) and stable disease (SD) are achieved from the start of cell infusion/the total number of evaluable cases (%).

CONTACTS AND LOCATIONS:
Overall Officials: Tingbo Liang, Principal Investigator — The First Affiliated Hospital, Zhejiang University
Locations (1):
- First affiliated hospital, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No